CLINICAL TRIAL: NCT06763224
Title: Prevalence of Neuropathic Pain After Non-instrumented Lumbar Spinal Surgery
Acronym: LomboDN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Colmar (Other)
Responsible Party: Sponsor
Other Study IDs: HCC-007; 2024-A00923-44 (Other: ID-RCB ANSM)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Disc Herniation; Lumbar Spinal Stenosis
Keywords: Neuropathic pain; Lumbar spinal surgery
MeSH Terms: conditions — Intervertebral Disc Displacement; Spinal Stenosis; Neuralgia | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire and Physical Exam — The neuropathic pain measured with the Neuropathic pain DN4 Questionnaire (Echelle de la Douleur Neuropathique en 4 questions - Neuropathic Pain Scale in 4 questions) The global pain measured with Visual Analogue Scale (VAS) The patient's permanent functional disability measured with the Oswestry disability index (ODI) The quality of life measured with the questionnaire EuroQol-5 Dimension (EQ-5D-5L)

SUMMARY:
Chronic neuropathic pain following lumbar spine surgery is often under-diagnosed and difficult to relieve. It can persist long after the operation, sometimes for months or even years, and has a major impact on the quality of life of patients who suffer from it. However, the scientific literature on the subject remains relatively poor, as evidenced by the absence of scientific studies on the prevalence of neuropathic pain after lumbar spinal surgery, whether instrumented or not.

The main aim of this study is to determine whether lumbar spine surgery has an impact on the prevalence of neuropathic pain. Participants will be followed up and complete a quality-of-life questionnaire for one year after surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients admitted for scheduled primary lumbar spine surgery without pedicle osteosynthesis or interbody cage.
* Pathology concerned by programmed surgery: herniated disc or lumbar spinal stenosis, uncomplicated by motor or sphincter deficits.
* Delay between 1st painful symptoms and surgery > 48h.

Non-inclusion criteria:

* Surgery scheduled within 48 hours of onset of symptoms.
* Presence of cauda equina syndrome
* Presence of motor-radicular deficit
* Patients with neurological pathology prior to surgery
* Major cognitive or sensory disorders preventing completion of the self-questionnaire
* Patients under guardianship
* Patients not covered by French social security.
* Patients who develop an identified neurological pathology after surgery, regardless of the initial surgery (e.g. multiple sclerosis, spinal cord injury, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Comparison of the proportion of patients with neuropathic pain between the day before surgery and 12 months after surgery. | The day before surgery and 12 months after surgery
  Comparison of the proportion of patients with a score ≥ 4 measured with the DN4 questionnaire one day before surgery and 12 months after surgery. The DN4 questionnaire (4-question neuropathic pain scale) is a diagnostic tool used to identify and assess neuropathic pain. The questionnaire aims to measure the presence of symptoms and signs commonly associated with neuropathic pain.
  The questionnaire comprises 10 items:
  * 7 items relate to the patient's description of his or her pain (burning, painful cold, electric shocks, tingling, numbness, itching).
  * 3 items are based on the clinician's sensory examination, focusing on touch and pinprick hypoesthesia, as well as brush-induced allodynia.
  The DN4 is scored out of 10 points. A score of 4 or more suggests the presence of neuropathic pain.

SECONDARY OUTCOMES:
Evolution of post-operative neuropathic pain | At 1, 3 and 6 months after surgery
  Proportion of patients with a DN4 score ≥ 4 at 1, 3 and 6 months post-operatively.
  The DN4 questionnaire (4-question neuropathic pain scale) is a diagnostic tool used to identify and assess neuropathic pain. The questionnaire aims to measure the presence of symptoms and signs commonly associated with neuropathic pain.
  The questionnaire comprises 10 items:
  * 7 items relate to the patient's description of his or her pain (burning, painful cold, electric shocks, tingling, numbness, itching).
  * 3 items are based on the clinician's sensory examination, focusing on touch and pinprick hypoesthesia, as well as brush-induced allodynia.
Evolution of overall pain | The day before surgery and at 1, 3, 6 and 12 months after surgery
  Global pain is measured using the Visual Analog Scale (VAS). The VAS is one of a number of pain assessment scales. Using a ruler, the score is determined by measuring the distance in mm on a 10 cm line between the "no pain" reference point and the patient's mark, giving a range of scores from 0 to 100. A higher score indicates greater pain intensity.
Evolution of functionality and disability of patients | The day before surgery and at 1, 3, 6 and 12 months after surgery
  The Oswestry Disability Index (ODI) is used to measure a patient's permanent functional disability. The ODI consists of 10 questions, scored from 0 to 5 (minimum to maximum). The total points for each section are added together, divided by the total possible points for all completed sections, and multiplied by 100 to create a disability percentage from 0 to 100%. A high percentage indicates significant disability.
Evolution of quality of life measured with EQ-5D-5L | The day before surgery and at 1, 3, 6 and 12 months after surgery
  The EuroQoL-5D-5L (EQ-5D-5L) self-administered questionnaire comprises 2 pages: one page with the 5-dimensional questionnaire EQ-5D and the visual analog quality-of-life scale EQ VAS. The EQ-5D explores the following 5 dimensions: mobility, personal care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, mild problems, moderate problems, severe problems and extreme problems. Patients are asked to indicate their state of health by ticking the box corresponding to the most appropriate statement in each of the five dimensions. The level chosen for each dimension corresponds to 1 number from 1 to 5 (1 = no problems, 5 = extreme problems).
  The VAS EQ records the patient's self-assessment of health status on a vertical visual analogue scale, the ends of which are entitled "The best health you can imagine" and "The worst health you can imagine". The VAS can be used as a quantitative measure of health status.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy VOIRIN, Principal Investigator — Centre Hospitalier de Colmar
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, France

IPD SHARING:
Plan to Share IPD: No